CLINICAL TRIAL: NCT01458288
Title: A Study to Evaluate the Safety, Pharmacokinetics, and Hematopoietic Stem Cell Mobilization of TG-0054 Alone or in Combination With G-CSF in Patients With Multiple Myeloma, Non-Hodgkin Lymphoma or Hodgkin Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GPCR Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG-0054-03
Record Dates: First submitted 2011-10-13; First posted 2011-10-24 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Multiple Myeloma; Non-hodgkin's Lymphoma; Hodgkin's Disease
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease

ARMS (1):
- TG-0054 (3.14 mg/kg) (Experimental): TG-0054 (3.14 mg/kg)
  Interventions: Drug: TG-0054

INTERVENTIONS:
Drug: TG-0054 — 3.14 mg/kg TG-0054 administrated via 15-min IV infusion(allow a maximum of four leukapheresis sessions)
  Other Names: burixafor

SUMMARY:
This Phase II study is to Evaluate the Safety, Pharmacokinetics, and Hematopoietic Stem Cell Mobilization of TG-0054 alone or in combination with G-CSF in Patients with Multiple Myeloma, Non-Hodgkin Lymphoma or Hodgkin Disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 75 years of age inclusive;
* Patients with confirmed pathology diagnosis of MM, NHL or HD;
* Potential candidate for autologous stem cell transplantation at Investigator's discretion;
* 4 weeks since last cycle of chemotherapy prior to the study drug administration;
* Total dose of melphalan received 200 mg in the most recent chemotherapy treatment;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Recovered from all acute toxic effects of prior chemotherapy at Investigator's discretion;
* White blood cell (WBC) count 3.0 x 109/L on screening laboratory assessments;
* Absolute neutrophil count 1.5 x 109/L on screening laboratory assessments;
* Platelet count 100 x 109/L on screening laboratory assessments;
* Serum creatinine 2.2 mg/dL on screening laboratory assessments;
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and total bilirubin < 2 x upper limit of normal (ULN) on screening laboratory assessments;
* Negative for human immunodeficiency virus (HIV);
* Adequate cardiac and pulmonary function to undergo leukapheresis at Investigator's discretion;
* For females, one of the following criteria must be fulfilled:

  1. At least one year post-menopausal, or
  2. Surgically sterile, or
  3. Willing to use a double-barrier method [intrauterine device (IUD) plus condom, spermicidal gel plus condom] of contraception from study Day 1 until 28 days after the last dose of TG-0054;
* Males must be willing to use a reliable form of contraception (use of a condom or a partner fulfilling the above criteria) from study Day 1 until 28 days after the last dose of TG-0054;
* Able to provide the signed informed consent.

Exclusion Criteria:

* Received radiation therapy to the pelvis;
* Received > 6 cycles of lenalidomide;
* Evidence of bone marrow involvement of lymphoma in NHL patients;
* Failed previous stem cell collection [failed to collect 2 x 106 CD34+ cells/kg within 4 leukapheresis sessions after receiving granulocyte colony-stimulating factor (G-CSF)];
* Patients who have undergone previous stem cell transplantation procedure;
* Received G-CSF within 2 weeks prior to the study drug administration;
* History of other cancer within the past 5 years excluding MM, NHL, HD, basal cell or squamous cell carcinoma of the skin;
* History of other hematologic disorders including bleeding or thromboembolic disease being treated with anti-coagulant;
* History of poor and uncontrollable cardiovascular or pulmonary disease such as myocardial infarction, cardiac arrhythmias, transient ischemic attack, stroke or Chronic Obstructive Pulmonary Disease (COPD) patients hospitalized more than two times a year due to underlying disease;
* Diagnosis of sickle cell anemia or documented sickle cell trait;
* Patients with proliferative retinopathy;
* Uncontrollable malignancy with MM, NHL or HD, or carcinomatous meningitis, at Investigator's discretion;
* Any infection required antibiotic treatment or unexplained fever above 38 °C within 3 days prior to dosing;
* Pregnant or breast-feeding;
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study;
* Received any other investigational drug within 1 month before entering the study;
* Received prior treatment with TG-0054 but withdrew early from this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W. Schuster, M.D., Principal Investigator — Stony Brook University Hospital
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Duration of the Study:
  This study will consist of a 14-day screening period, a 2- to 11-day treatment period, and a 7-day follow-up period.
  Number of Patients:
  Approximately 12 treatment evaluable patients will be enrolled in this study.
  Study Location: Single site in US.
Groups:
- TG-0054 (3.14 mg/kg TG-0054 Administrated Via 15-min IV Infus): TG-0054 (3.14 mg/kg)
  TG-0054: 3.14 mg/kg TG-0054 administrated via 15-min IV infusion(allow a maximum of four leukapheresis sessions)
Period: Overall Study
Arm/Group | TG-0054 (3.14 mg/kg TG-0054 Administrated Via 15-min IV Infus)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- TG-0054 (3.14 mg/kg Administrated Via 15-min IV Infusion): TG-0054 (3.14 mg/kg)
  TG-0054: 3.14 mg/kg TG-0054 administrated via 15-min IV infusion(allow a maximum of four leukapheresis sessions)
Arm/Group | TG-0054 (3.14 mg/kg Administrated Via 15-min IV Infusion)
Number analyzed (Participants) | 12
Age, Customized [Number; unit: participants]
  18 to 75 years old | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving the CD34+ Hematopoietic Stem Cell (HSC) Mobilization Target of ≧2.5×1000000 Cells/kg
Description: Patients were all with multiple myeloma (MM), Non-Hodgkin lymphoma (NHL) or Hodgkin disease (HD).
  Number of patients who mobilized the targeted total number of CD34+ cells within a maximum of 4 leukapheresis sessions in study arm 1 and arm 3. Patients in arm 1 followed administration of TG-0054 (3.14 mg/kg) alone and leukapheresis start from study day 1. Patients in arm 3 followed administration of TG-0054 (3.14 mg/kg) combined with granulocyte colony-stimulating factor (G-CSF) and leukapheresis start from study day 8.
Time Frame: 1 week
Measure: Number; unit: participants
Groups:
- TG-0054 (3.14 mg/kg): Patients followed administration of TG-0054 (3.14 mg/kg) alone and leukapheresis start from study day 1.
- TG-0054 (3.14 mg/kg)+G-CSF: Patients followed administration of TG-0054 (3.14 mg/kg) combined with granulocyte colony-stimulating factor (G-CSF) and leukapheresis start from study day 8.
Arm/Group | TG-0054 (3.14 mg/kg) | TG-0054 (3.14 mg/kg)+G-CSF
Number analyzed (Participants) | 7 | 5
participants | 7 | 5

2. Secondary Outcome: the Average Number of Leukapheresis Sessions
Description: To determine the average number of leukapheresis sessions required to collect 2.5 x10^6 CD34+ cells/kg.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: number of leukapheresis sessions
Arm/Group | TG-0054 (3.14 mg/kg) | TG-0054 (3.14 mg/kg)+G-CSF
Number analyzed (Participants) | 7 | 5
number of leukapheresis sessions | 2.0 (0.82) | 1.4 (0.55)

3. Secondary Outcome: Circulating CD34+ Cell Count in Peripheral Blood
Description: Calculate the median total CD34+ cell counts across all leukapheresis sessions following TG 0054 administration alone and in combination with G-CSF mobilization in order to evaluate the pharmacodynamics (PD) of TG-0054 by determining circulating CD34+ cell counts in peripheral blood.
Time Frame: pre-dose(-2 to 0 h),2, 4 and 6 hr after dosing.
Measure: Median (Full Range); unit: cells/kg
Arm/Group | TG-0054 (3.14 mg/kg) | TG-0054 (3.14 mg/kg)+G-CSF
Number analyzed (Participants) | 7 | 5
cells/kg | 6000000 [4000000 to 10000000] | 5000000 [4000000 to 21000000]

ADVERSE EVENTS:
Time Frame: 9 months, from 23-Oct-2012 to 09-Jul-2013
Arm/Group | TG-0054 (3.14 mg/kg Administrated Via 15-min IV Infusion)
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 10/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TG-0054 (3.14 mg/kg Administrated Via 15-min IV Infusion) (N=12)
Diarrhoea (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Paraesthesia oral (Gastrointestinal disorders) | 2
Blood pressure increased (Investigations) | 2
Haemoglobin decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Neuropathy peripheral (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Chest discomfort (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days